CLINICAL TRIAL: NCT00001128
Title: A Pilot, Proof-of-Concept, Dose-Escalating Trial of Recombinant Human Interleukin-12 (rhIL-12) Versus Placebo Along With Paromomycin and Azithromycin for Chronic Cryptosporidiosis in AIDS
Brief Title: Treatment of Chronic Cryptosporidiosis in AIDS Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genetics Institute (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: DAIDS R001
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2003-06

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Cryptosporidiosis; Acquired Immunodeficiency Syndrome; Azithromycin; Paromomycin; Interleukin-12
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Interleukin-12; Paromomycin; Azithromycin

INTERVENTIONS:
Drug: Interleukin-12
Drug: Paromomycin sulfate
Drug: Azithromycin

SUMMARY:
The purpose of this study is to see if it is safe and effective to add interleukin-12 (IL-12) to the standard drug combination (paromomycin plus azithromycin) used to treat cryptosporidiosis in AIDS patients. Doctors would like to find out if the combination of IL-12, paromomycin, and azithromycin is more effective than paromomycin and azithromycin alone.

Cryptosporidiosis is a type of opportunistic (AIDS-related) infection seen in HIV-positive patients as their immune systems weaken. It is caused by a parasite that invades the intestinal tract, and it can cause watery diarrhea, stomach cramps, an upset stomach, or a fever. Antibiotics (paromomycin and azithromycin) are usually used to treat cryptosporidiosis. In this study, doctors will look at the effectiveness of using IL-12. IL-12 is a type of protein naturally produced by certain types of cells of the immune system and is believed to be important for immune function. Doctors hope that IL-12 can help boost the immune system in fighting cryptosporidiosis.

DETAILED DESCRIPTION:
Cryptosporidium parvum, an intracellular protozoan parasite, is a frequent cause of chronic diarrhea in HIV-infected patients, causing significant morbidity and mortality. Highly effective antiparasitic treatment for this infection is not currently available. Paromomycin and azithromycin have some efficacy and have been used in combination in a small number of patients. Immune reconstitution with highly active antiretroviral therapy appears to be the most effective therapy, but this is not possible for all patients. Interferon gamma expression is strongly associated with control of cryptosporidiosis, and IL-12 is the cytokine primarily responsible for stimulation of interferon gamma expression in vivo. It is hoped that treatment with recombinant human IL-12 can result in stimulation of an intestinal cytokine response in AIDS patients with cryptosporidiosis and that response combined with chemotherapy can lead to the elimination of detectable numbers of Cryptosporidium oocysts from the stools.

All patients receive azithromycin and paromomycin, and patients are randomized to add either IL-12 or placebo. IL-12 (or placebo) injections are given twice a week. Patients take their study medications for 4 weeks. During this time, they will be asked to record bowel movements and any symptoms they experience. Patients return to the clinic at least twice a week to receive IL-12 (or placebo) injections. At Weeks 2 and 4, patients are seen by one of the principal investigators. Blood samples are obtained for viral load measurements and CD4 count, as well as routine urinalysis. Patients undergo upper endoscopy with jejunal biopsy and colonoscopy with ileal biopsy between Weeks 2 and 4 of therapy for assays of intestinal cytokine expression. A final clinic visit occurs 12 weeks post-therapy for a physical exam and blood tests.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count below 150 cells/mm3.
* Have been on stable anti-HIV therapy that includes at least 2 nucleoside analogues for at least 4 weeks.
* Have chronic diarrhea (3 bowel movements a day that are loose or watery, for 5 days per week over 3 weeks).
* Test positively for Cryptosporidium.
* Are at least 18 years old.
* Agree to use effective methods of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have any other active opportunistic (AIDS-related) infection.
* Require intravenous (IV) fluids.
* Have a history of an allergy to certain medications, such as colony-stimulating factors (G-CSF or GM-CSF) or a type of antibiotic.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Clinton White, Principal Investigator
Locations (1):
- Pablo C. Okhuysen, Houston, Texas, United States